CLINICAL TRIAL: NCT03005834
Title: Incidence of Cancers in Patients With Atherosclerotic Cardiovascular Diseases
Brief Title: The Sakakibara Health Integrative Profile Cohort Study
Acronym: SHIP-CS
Status: Completed | Type: Observational
Sponsor: Sakakibara Heart Institute (Other)
Responsible Party: Principal Investigator, Makoto Suzuki, Principal Investigator, Department of Cardiology, Sakakibara Heart Institute
Other Study IDs: SHIP01
Record Dates: First submitted 2016-12-26; First posted 2016-12-29 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Cancer
Keywords: Atherosclerotic cardiovascular diseases, cancers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1020 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atherosclerotic CVD: Atherosclerotic cardiovascular diseases (CVD) included coronary artery diseases, aortic diseases and peripheral artery diseases.
  Interventions: Other: incidence of cancers
- Non-atherosclerotic CVD: Non-atherosclerotic cardiovascular diseases (CVD) were any CVD except atherosclerotic CVD and congenital CVD.
  Interventions: Other: incidence of cancers

INTERVENTIONS:
Other: incidence of cancers — With a continuous surveillance system to track all subsequent incidents of CVD and/or non-CVD via direct contact in the outpatient department, hospital records, and a mailed questionnaire at least once a year, an incidence of cancers was identified.

SUMMARY:
Because of the genetic and traditional commonalities between the underlying causes of atherosclerotic cardiovascular diseases (CVD) and cancers, we hypothesized that patients with atherosclerotic CVD may have a high incidence of cancers when compared with those with non-atherosclerotic CVD. To address this hypothesis, we investigated longitudinal clinical outcomes in a total of 32,095 consecutive patients with CVD enrolled in the Sakakibara Health Integrative Profile (SHIP) cohort study which was launched in 2006 for the purpose of improving healthy life expectancy in patients with CVD in our institute.

DETAILED DESCRIPTION:
The SHIP cohort study was launched in 2006 for the purpose of improving healthy life expectancy in patients with any cardiovascular diseases (CVD) who were admitted to the Sakakibara Heart Institute. The study used a continuous surveillance system to track all subsequent incidents of CVD and/or non-CVD including cancers, via direct contact in the outpatient department, hospital records, and a mailed questionnaire at least once a year. Organ sites of cancers were also identified whenever possible. The study sorted any diagnoses of CVD into nine categories, namely coronary artery diseases, aortic diseases, peripheral artery diseases, myocardial diseases, unclassified or any-cause heart failure, valvular heart diseases, arrhythmias, congenital CVD, and others. For example, if a patient had a couple of diseases, he or she had a plural category. Cerebrovascular diseases were included in the category of 'others' because of the mixed cause for the diseases such as embolic strokes, lacunar infarction, cardio-embolic strokes, and hemorrhagic strokes, etc. Atherosclerotic CVD were defined by the presence of one or more of the following three diseases: coronary artery diseases, aortic diseases and peripheral artery diseases. With regard to the detail of coronary artery diseases, there were acute coronary syndromes, previous myocardial infarction and stable ischemic heart diseases. Aortic diseases consisted of acute aortic syndromes and aortic aneurysms. Non-atherosclerotic CVD were defined as any CVD except atherosclerotic and congenital CVD. The SHIP cohort study also handled to define lifestyle related diseases when confirmed a diagnosis of one or more of the presence of hypertension, dyslipidemia, diabetes mellitus and chronic kidney disease in accordance with the universal criteria. A history of tobacco smoking was also identified. Among a total of 36,151 patients with any CVD enrolled in the SHIP cohort study between June 2006 and July 2014, we excluded 245 patients who had already been diagnosed with any cancers at the time of enrollment in the SHIP cohort study, and 3,811 patients with congenital CVD including Marfan syndrome. Thus, we analyzed a total of 32,095 consecutive patients with acquired CVD in the present study.Our study was conducted in two steps to assess an incidence of cancers in patients with acquired CVD. The first step consisted of a comparison between those with atherosclerotic CVD and non-atherosclerotic CVD with regard to an incidence of cancers. The second step determined the association between a singular presence versus a plural presence of atherosclerotic CVD and an incidence of cancers.

ELIGIBILITY:
Inclusion Criteria:

* Among a total of 36,151 patients with any CVD enrolled in the SHIP cohort study between June 2006 and July 2014, we analyzed a total of 32,095 consecutive patients with acquired CVD in the present study after excluding 4,056 patients with known cancers and/or congenital CVD.

Exclusion Criteria:

* We excluded 245 patients who had already been diagnosed with any cancers at the time of enrollment in the SHIP cohort study, and 3,811 patients with congenital CVD including Marfan syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 36,151 patients (58% male, 61±23 years) with any cardiovascular diseases (CVD) enrolled in the SHIP cohort study between June 2006 and July 2014.
Sampling Method: Non-Probability Sample
Enrollment: 32095 (Actual)
Dates: Start 2006-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
incidence of cancers | July, 2014

SECONDARY OUTCOMES:
any cause mortality | July, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Suzuki, MD, Principal Investigator — Sakakibara Heart Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suzuki M, Tomoike H, Sumiyoshi T, Nagatomo Y, Hosoda T, Nagayama M, Ishikawa Y, Sawa T, Iimuro S, Yoshikawa T, Hosoda S. Incidence of cancers in patients with atherosclerotic cardiovascular diseases. Int J Cardiol Heart Vasc. 2017 Sep 14;17:11-16. doi: 10.1016/j.ijcha.2017.08.004. eCollection 2017 Dec. PMID 28948207